CLINICAL TRIAL: NCT01923636
Title: Evaluation of the Prognostic Value of Clinical, Imaging, Immunological and Virological Markers in the Neonatal Period for the Development of Neurosensorial Sequelae at 1 Year in Children Infected by Cytomegalovirus in Utero.
Brief Title: Prognostic Value of Neonatal Markers for the Development of Neurosensorial Sequelae in Children Infected by Cytomegalovirus in Utero
Acronym: CYMEPEDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120114; AOM12196
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Cytomegalovirus, congenital, handicap
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- detection of CMV (Other): Cohort of neonates less than 1 month with congenital CMV infection at birth objectified by the detection of CMV in a urine sample, in saliva or blood (fresh or Guthrie card) obtained in the first 10 days life
  Interventions: Other: detection of CMV

INTERVENTIONS:
Other: detection of CMV — Clinical, radiological and laboratory (virological and immunological) standardized reports

SUMMARY:
The main objective of this study is to validate , in the neonatal period, a prognostic score for the development of neurosensorineural sequelae at 1 year and at 2 years in neonates infected in utero by cytomegalovirus. This score will be based on clinical, imaging and biological criteria .

The second objective of the study is to estimate the prevalence of this infection in France and to describe its epidemiology through the screening of 12,000 consecutive neonates.

DETAILED DESCRIPTION:
Infection with cytomegalovirus (CMV) is the most frequent cause of congenital neurological handicap of infectious origin in industrialized countries. Around 10% of infected neonates have symptoms and more than 50% of those will develop long term neurological sequelae and sensorineural hearing loss. Among asymptomatic infected neonates 10 to 15% will ultimately develop hearing loss. To establish the prognosis of infected neonates remains difficult and the purpose of the study is to better define early prognosis factors The true burden of CMV congenital infection is unknown in France: the prevalence of the infection as well as the description of its epidemiology (proportion of symptomatic and asymptomatic cases, rate of long term sequelae, proportion of cases following primary or secondary maternal infections) are unknown.

ELIGIBILITY:
Inclusion Criteria:

Main objective: Neonate less than 1 month with congenital CMV infection at birth objectified by the detection of CMV in a urine sample, in saliva or blood (fresh or Guthrie card) obtained in the first 10 days life

* Whose parents accept regular monitoring by the paediatrician investigator
* For which a medical examination has been made
* Affiliated with a social security system
* And whose mother has given its written consent to the participation of their child to study

Exclusion Criteria:

- Children participating in an interventional study

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Prognostic value of neonatal markers (clinical, imaging and biological) for the development of neurosensorial sequelae at 1 year of age | One year
  Assessment will include standardised clinical evaluation, cerebral ultrasound, cerebral MRI, audiometric tests, developmental tests, virological tests (viral load in blood and saliva) and immunological tests (cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), Natural Killer (NK) and cytokines).

SECONDARY OUTCOMES:
to evaluate the prevalence of congenital CMV in France: | At birth
  screening by CMV PCR in a saliva sample collected in delivery room will be proposed to all mothers with a live birth neonate born in the Necker or Poissy
Prognosis value of antenatal imaging | one year
  To compare neurodevelopmental and sensorineural sequelae at one year with the result of antenatal imaging (ultrasound and MRI)
Prognostic value of the periodic measurement of the kinetics of viral load shedding | One year
  To evaluate the prognostic value of the kinetics of CMV viral load in blood and in saliva from birth to 1 year old for the occurrence of neurodevelopmental and sensorineural sequelae
neurodevelopmental and sensorineural sequelae according to the type of maternal infectionsequelae | One year
  Compare the proportion of neurodevelopmental and sensorineural sequelae according to the type of maternal infection (primary or secondary).
Prevalence and description of congenital CMV infection in 10,000 French neonates | 1 week
  Screening of congenital CMV infection in a population of 10,000 consecutive newborns in 2 French maternities

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Bussieres, MD, Study Director — APHP
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Fourgeaud J, Magny JF, Couderc S, Garcia P, Maillotte AM, Benard M, Pinquier D, Minodier P, Astruc D, Patural H, Ugolin M, Parat S, Guillois B, Garenne A, Guilleminot T, Parodi M, Bussieres L, Ville Y, Leruez-Ville M. Clinical Value of Serial Quantitative Analysis of Cytomegalovirus DNA in Blood and Saliva Over the First 24 Months of Life in Congenital Infection: The French Cymepedia Cohort. J Pediatr. 2023 Feb;253:197-204.e5. doi: 10.1016/j.jpeds.2022.09.040. Epub 2022 Sep 28. PMID 36181870
- [Background] Leruez-Ville M, Ren S, Magny JF, Jacquemard F, Couderc S, Garcia P, Maillotte AM, Benard M, Pinquier D, Minodier P, Astruc D, Patural H, Ugolin M, Parat S, Guillois B, Garenne A, Parodi M, Bussieres L, Stirnemann J, Sonigo P, Millischer AE, Ville Y. Accuracy of prenatal ultrasound screening to identify fetuses infected by cytomegalovirus which will develop severe long-term sequelae. Ultrasound Obstet Gynecol. 2021 Jan;57(1):97-104. doi: 10.1002/uog.22056. PMID 32339337
- [Background] Faure-Bardon V, Magny JF, Parodi M, Couderc S, Garcia P, Maillotte AM, Benard M, Pinquier D, Astruc D, Patural H, Pladys P, Parat S, Guillois B, Garenne A, Bussieres L, Guilleminot T, Stirnemann J, Ghout I, Ville Y, Leruez-Ville M. Sequelae of Congenital Cytomegalovirus Following Maternal Primary Infections Are Limited to Those Acquired in the First Trimester of Pregnancy. Clin Infect Dis. 2019 Oct 15;69(9):1526-1532. doi: 10.1093/cid/ciy1128. PMID 30596974
- [Background] Leruez-Ville M, Magny JF, Couderc S, Pichon C, Parodi M, Bussieres L, Guilleminot T, Ghout I, Ville Y. Risk Factors for Congenital Cytomegalovirus Infection Following Primary and Nonprimary Maternal Infection: A Prospective Neonatal Screening Study Using Polymerase Chain Reaction in Saliva. Clin Infect Dis. 2017 Aug 1;65(3):398-404. doi: 10.1093/cid/cix337. PMID 28419213